CLINICAL TRIAL: NCT01094873
Title: A Phase I Study to Assess the Safety and Immunogenicity of Ad6NSmut and AdCh3NSmut in Patients With Hepatitis C Virus Infection
Brief Title: Study of a Novel Therapeutic Vaccine for Hepatitis C Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReiThera Srl (Industry)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV002TV; 2008-006127-32 (EudraCT Number); GTAC162 (Other: Gene Therapy Advisory Committee (GTAC), UK)
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; HCV; Adenovirus; Vaccine
MeSH Terms: conditions — Hepatitis C; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Arm A, group 1 (Experimental): Interventions: AdCh3NSmut; Ad6NSmut. Administration schedule: 1 dose AdCh3NSmut 5 x 10^8vp at week 14 and 1 dose Ad6NSmut 5 x 10^8vp at week 24, after starting PEG-IFN and ribavirin therapy.
  Patients: 2
  Interventions: Biological: AdCh3NSmut; Biological: Ad6NSmut
- Arm A, group 2 (Experimental): Interventions: AdCh3NSmut; Ad6NSmut. Administration schedule: 1 dose AdCh3NSmut 5 x 10^9vp at week 14 and 1 dose Ad6NSmut 5 x 10^9vp at week 24, after starting PEG-IFN and ribavirin therapy.
  Patients: 2
  Interventions: Biological: AdCh3NSmut; Biological: Ad6NSmut
- Arm A, group 3 (Experimental): Interventions: AdCh3NSmut; Ad6NSmut. Administration schedule: 1 dose AdCh3NSmut 2.5 x 10^10vp at week 14 and 1 dose Ad6NSmut 2.5 x 10^10vp at week 24, after starting PEG-IFN and ribavirin therapy.
  Patients: 6
  Interventions: Biological: AdCh3NSmut; Biological: Ad6NSmut
- Arm A, group 4 (Experimental): Interventions: AdCh3NSmut; Ad6NSmut. Administration schedule: 1 dose AdCh3NSmut 2.5 x 10^10vp at week 2 and 1 dose Ad6NSmut 2.5 x 10^10vp at week 12, after starting PEG-IFN and ribavirin therapy.
  Patients: 6
  Interventions: Biological: AdCh3NSmut; Biological: Ad6NSmut
- Arm A, group 5 (Experimental): Interventions: AdCh3NSmut; Ad6NSmut. Administration schedule: 1 dose AdCh3NSmut 2.5 x 10^10vp at weeks 14 and 18, and 1 dose Ad6NSmut 2.5 x 10^10vp at week 28, after starting PEG-IFN and ribavirin therapy.
  Patients: 4
  Interventions: Biological: AdCh3NSmut; Biological: Ad6NSmut
- Arm A, group 6 (Experimental): Interventions: AdCh3NSmut; Ad6NSmut. Administration schedule: 1 dose AdCh3NSmut 2.5 x 10^10vp at weeks 2 and 6, and 1 dose Ad6NSmut 2.5 x 10^10vp at week 16, after starting PEG-IFN and ribavirin therapy.
  Patients: 4
  Interventions: Biological: AdCh3NSmut; Biological: Ad6NSmut
- Arm B, group 1 (Experimental): Interventions: AdCh3NSmut; Ad6NSmut. Administration schedule: 1 dose AdCh3NSmut 5 x 10^8vp at week 4 and 1 dose Ad6NSmut 5 x 10^8vp at week 14.
  Patients: 2
  Interventions: Biological: AdCh3NSmut; Biological: Ad6NSmut
- Arm B, group 2 (Experimental): Interventions: AdCh3NSmut; Ad6NSmut. Administration schedule: 1 dose AdCh3NSmut 5 x 10^9vp at week 4 and 1 dose Ad6NSmut 5 x 10^9vp at week 14.
  Patients: 2
  Interventions: Biological: AdCh3NSmut; Biological: Ad6NSmut
- Arm B, group 3 (Experimental): Interventions: AdCh3NSmut; Ad6NSmut.
  1 dose AdCh3NSmut 2.5 x 10^10vp at week 4 and 1 dose Ad6NSmut 2.5 x 10^10vp at week 14.
  Patients: 4
  Interventions: Biological: AdCh3NSmut; Biological: Ad6NSmut

INTERVENTIONS:
Biological: AdCh3NSmut — Genetic vaccines against Hepatitis C virus infection
Biological: Ad6NSmut — Genetic vaccine against Hepatitis C virus infection

SUMMARY:
HCV002TV is a Phase I study to ascertain the safety and immunogenicity of a novel vaccine against Hepatitis C virus (HCV) in chronically infected patients. The vaccine is based on the sequential delivery, by intramuscular route, of two different adenoviral vectors, of chimpanzee and human origin respectively, bearing the same genetic information for HCV antigens (NS region).

The two recombinant vaccine vectors, called AdCh3NSmut and Ad6NSmut, are weakened and unable to multiply within the body; they are designed to induce an immune response against HCV proteins. AdCh3NSmut and Ad6NSmut are being used in the ongoing HCV001 study in healthy volunteers with very good safety and immunogenicity results.

HCV002TV is a dose-escalation study; the AdCh3NSmut is administered as priming vaccination and Ad6NSmut as boosting vaccination.

The trial includes:

* Arm A, in which vaccinated patients are into Interferon-ribavirin therapy (the gold standard therapy for hepatitis C);
* Arm B, in which vaccinated patients are not into therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient must satisfy all the following criteria to be eligible for the study:

  * HCV infected with genotype-1 infection
  * Adults aged 18 to 65 years (inclusive)
  * In arms A1-A3 patients will only be vaccinated if they have a >2log drop in viral load at week 12 of IFN-alpha and ribavirin therapy. Vaccination will then occur at week 14 into IFN-alpha and ribavirin therapy.
  * Resident in or near the trial sites for the duration of the vaccination study
  * Able and willing (in the Investigator's opinion) to comply with all study requirements
  * For women of child bearing potential, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of vaccination
  * For men to use barrier contraception until three months after the last vaccination
  * Written informed consent

Exclusion Criteria:

* The patient may not enter the study if any of the following apply:

  * Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
  * Prior receipt of a recombinant simian or human adenoviral vaccine
  * Clinical, biochemical, ultrasonographic, or liver biopsy (histology) evidence of cirrhosis or portal hypertension
  * Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
  * Patients likely to have been infected with HCV within the last 12 months
  * History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g., Kathon
  * Patients who failed to respond (non-responders) to previous IFN-alpha monotherapy
  * Patients who received IFN-alpha and ribavirin in the past and who were non-responders or relapsed during or after therapy
  * History of clinically significant contact dermatitis
  * For Arm A, patients must be treatment naïve (i.e. never have had previous IFNα or ribavirin treatment). Arm B may include patients who have previously been treated for HCV and failed to achieve a sustained virological response (defined by undetectable HCV by PCR at 6 months post cessation of treatment)
  * Any history of anaphylaxis in reaction to vaccination
  * Pregnancy, lactation or willingness/intention to become pregnant during the study
  * History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
  * Any other serious chronic illness requiring hospital specialist supervision
  * Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
  * Current suspected or known injecting drug abuse
  * Seropositive for hepatitis B surface antigen (HBsAg)
  * Seropositive for HIV (antibodies to HIV) at screening
  * Seropositive for simian adenovirus 3 (antibodies to AdCh3) at titres >200, at screening
  * Seropositive for human adenovirus 6 (antibodies to Ad6) at titres >200, at screening
  * Any other significant disease, disorder or finding, which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or may influence the result of the study, or the patient's ability to participate in the study
  * Any other finding which in the opinion of the investigators would significantly increase the risk of having an adverse outcome from participating in the protocol
  * Individuals who have had a temperature >38°C in the 3 days preceding vaccination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety and immunogenicity | Different time points depending on the study groups with a 6-months follow-up after last vaccination for all groups
  To assess the safety and immunogenicity of new hepatitis C vaccine candidates, AdCh3NSmut and Ad6NSmut when administered in a prime/boost regimen to HCV infected patients. The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events. The specific endpoint of cellular immune response will be collected via IFN-gamma ELISpot assay and other exploratory immunological tests.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Barnes, MD, Study Chair — University of Oxford, UK; David Mutimer, Dr., Principal Investigator — University of Birmingham
Locations (2):
- United Kingdom (2):
  - Wellcome Clinical Research Facility, Queen Elizabeth's Hospital, University Hospital Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - John Radcliffe Hospital, Headley Way, Headington, Oxford

REFERENCES:
- See also: HCV002TV study sponsor Web site — http://www.okairos.com